CLINICAL TRIAL: NCT03039842
Title: Combination of Dextromethorphan and Memantine in Treating Bipolar Disorder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ru-Band Lu, Distinguished Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CombindBP2014
Record Dates: First submitted 2014-08-29; First posted 2017-02-01 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Bipolar Disorder II
Keywords: dextromethorphan; memantine; treatment response
MeSH Terms: conditions — Bipolar Disorder | interventions — Dextromethorphan; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 30 mg DM (Experimental): 30mg dextromethorphan+valproate
  Interventions: Drug: Dextromethorphan
- 5 mg MM (Experimental): 5mg memantine+valproate
  Interventions: Drug: Memantine
- DM+MM (Experimental): dextromethorphan+memantine+ valproate
  Interventions: Drug: dextromethorphan+memantine
- placebo (Placebo Comparator): Placebo+valproate
  Interventions: Drug: placebo+valproate

INTERVENTIONS:
Drug: Dextromethorphan
  Other Names: 30mg dextromethorphan
  Arms: 30 mg DM
Drug: Memantine
  Other Names: 5mg memantine+valproate
  Arms: 5 mg MM
Drug: dextromethorphan+memantine
  Arms: DM+MM
Drug: placebo+valproate
  Arms: placebo

SUMMARY:
This is a research clinical trial of double-blind, stratified randomized, parallel group, two-centre study. It will be conducted in a total of 250~300 male and female subjects from the Department of Psychiatry at National Cheng Kung University Hospital. Eligible subjects will be psychiatric out- and in-patients, aged between 18~65 years old, who have psychiatric evaluation with clinically suspected of having bipolar II disorder and fulfill the inclusion and exclusion criteria. The add-on double-blind study treatment with dextromethorphan/place will commence at randomization for while patients continue open-label valproate. Subjects will be enrolled for 12 weeks double-blind add-on treatment and randomly assigned to (1) 30mg dextromethorphan+valproate, (2) 5mg memantine+valproate, (3) dextromethorphan+memantine+valproate or (4) placebo+valproate. Concomitant benzodiazepine medication (preferably up to 8mg lorazepam) may be used for daytime sedation, agitation or insomnia during the study. For the consideration of the less influence to immune-system, resperidone 1-3mg/daily and fluoxetine maximum 20mg/daily will be chose. We will measure the treatment response and side effect to clarify the curative effect of DM and memantine add-on therapy to valproate in the treatment of bipolar disorders. This study is being performed to investigate the possibly significant beneficial effects on the subtypes of bipolar disorders psychopathology.

DETAILED DESCRIPTION:
A total of 250~300 male and female subjects from the Department of Psychiatry at National Cheng Kung University Hospital. Eligible subjects who are aged between 18~65 years old and clinically suspected of having bipolar II disorder are invited. The add-on double-blind study treatment with dextromethorphan/place will commence at randomization for while patients continue open-label valproate. Subjects will be enrolled for 12 weeks double-blind add-on treatment and randomly assigned to (1) 30mg dextromethorphan+valproate, (2) 5mg memantine+valproate, (3) dextromethorphan+memantine+valproate or (4) placebo+valproate. Concomitant benzodiazepine medication (preferably up to 8mg lorazepam) may be used for daytime sedation, agitation or insomnia during the study. For the consideration of the less influence to immune-system, resperidone 1-3mg/daily and fluoxetine maximum 20mg/daily will be chose. We will measure the treatment response and side effect to clarify the curative effect of DM and memantine add-on therapy to valproate in the treatment of bipolar disorders. This study is being performed to investigate the possibly significant beneficial effects on the subtypes of bipolar disorders psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* A 2-day minimum for hypomania to diagnose bipolar II disorder
* A total of Hamilton Rating Scale for Depression scored at least 18 or Young Mania Rating Scale scored at least 14 at the screening stage
* Must allow to ensure acceptable compliance and visit

Exclusion Criteria:

* Pregnant females or nursing
* Women of childbearing potential not using adequate contraception
* Received dextromethorphan, memantine, other antiinflammatory medication within 1 week prior
* Clinically significant medical condition (cardiac, hepatic and renal disease)
* Received electroconvulsive therapy patients within 4 weeks prior to the first dose of double-blind medication
* Increase in total SGOT, SGPT, BUN and creatinine by more than 3X upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
treatment change assessed by plasma levels of cytokines (e.g., IL-6, IL-8) | baseline, week 1, week 2, week 4, week 8, week 12
  change assessment

SECONDARY OUTCOMES:
depression change change | baseline, week 1, week 2, week 4, week 8, week 12
  depression change assessed by Hamilton Depression Rating Scale
manic state change | baseline, week 1, week 2, week 4, week 8, week 12
  Manic symptom assessed by Young Mania Rating Scale

OTHER OUTCOMES:
attention function change | baseline, week 12
  attention change assessed by CPT
memory change | baseline, week 12
  memory change assessed by WMS
executive functioning change | baseline, week 12
  executive function change assessed by WCST

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Band Lu, MD, Principal Investigator — Department of Psychiatry, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee SY, Wang TY, Chen SL, Chang YH, Chen PS, Huang SY, Tzeng NS, Wang LJ, Lee IH, Chen KC, Yang YK, Hong JS, Lu RB. Combination of dextromethorphan and memantine in treating bipolar spectrum disorder: a 12-week double-blind randomized clinical trial. Int J Bipolar Disord. 2020 Mar 2;8(1):11. doi: 10.1186/s40345-019-0174-8. PMID 32115672